CLINICAL TRIAL: NCT07348653
Title: A Phase I Study of Safety, Tolerability, Pharmacokinetics and Efficacy of MG2512 Injection in Participants With Advanced Solid Tumors
Brief Title: A Study of MG2512 Injection in Participants With Advanced Solid Tumors
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Mabgen Biopharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MG2512-101
Record Dates: First submitted 2026-01-08; First posted 2026-01-16 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MG2512 Injection Group (Experimental)
  Interventions: Drug: MG2512 Injection

INTERVENTIONS:
Drug: MG2512 Injection — MG2512 injection.

SUMMARY:
This is an open-label, multi-center, multiple dose Phase 1 study to evaluate the safety, tolerability, pharmacokinetics and efficacy of MG2512 injection in participants with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary participation and written informed consent.
2. 18-75 years old, no gender limitation.
3. Eastern Cooperative Oncology Group (ECOG) score: 0-1.
4. With a life expectancy ≥ 3 months.
5. Patients with recurrent or metastatic solid tumors that have been histologically or cytologically confirmed to be incurable through surgery or radical radiotherapy and chemotherapy, who have experienced disease progression after standard treatment, or have no standard treatment plan, or are not suitable for standard treatment.
6. Be able to provide fresh or archived tumour tissue.
7. At least one measurable lesion according to RECIST v1.1.
8. Adequate bone marrow reserve and organ function.
9. Contraception is required during the trial.

Exclusion Criteria:

1. Meningeal metastasis history or clinical symptoms of central nervous system metastasis.
2. History of other malignant tumors within 5 years before the first use of the study drug.
3. Uncontrollable tumor-related pain or symptomatic hypercalcemia.
4. Having severe cardiovascular and cerebrovascular diseases.
5. Presence of bleeding symptoms with significant clinical significance within 3 months before the first use of the study drug.
6. Uncontrollable effusion within 2 weeks before the first use of the study drug.
7. Subjects with history of interstitial pneumonia or lung diseases that severely affect lung function.
8. Having a severe infection within 4 weeks before the start of study treatment.
9. History of immunodeficiency, including positive HIV test results; presence of active hepatitis B.
10. Subjects with active pulmonary tuberculosis infection within 1 year before enrollment.
11. Adverse reactions from previous antitumor treatment that have not recovered to CTCAE ≤ Grade 1.
12. Failure to meet the following requirements for previous treatment washout: receipt of anti-tumor treatments such as chemotherapy, biological therapy, targeted therapy, immunotherapy, or other non-marketed investigational drug treatments within 4 weeks before the first use of the study drug.
13. Receipt of chest radiotherapy with a dose > 30 Gy within 24 weeks before the first use of the study drug.
14. Subjects with previous or planned allogeneic bone marrow transplantation or solid organ transplantation.
15. Subjects with known allergy to any component or excipient of the MG2512 product.
16. Subjects with other factors that may affect the study results or lead to forced premature termination of the study, as judged by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) | 3 weeks.
Maximum tolerated dose (MTD) | 3 weeks.
Recommended Phase 2 Dose (RP2D) | From screening period up to study completion, an average of 1 year.
Adverse events (AEs) | From screening period up to study completion, an average of 1 year.

SECONDARY OUTCOMES:
Blood concentration of MG2512 after single and continuous administration | From screening period up to study completion, an average of 1 year.
Time to reach maximum plasma concentration (Tmax) | From screening period up to study completion, an average of 1 year.
  PK parameters of MG2512 after single and continuous administration.
Maximum plasma Concentration (Cmax) | From screening period up to study completion, an average of 1 year.
  Pharmacokinetics (PK) parameters of MG2512 after single and continuous administration.
Area under the curve from zero to time t (AUC0-t) | From screening period up to study completion, an average of 1 year.
  Pharmacokinetics (PK) parameters of MG2512 after single and continuous administration.
Drug Resistant Antibody (ADA) to MG2512 | From screening period up to study completion, an average of 1 year.
Objective response rate (ORR) | From screening period up to study completion, an average of 1 year.
Disease control rate (DCR) | From screening period up to study completion, an average of 1 year.
Progression-free survival (PFS) | From screening period up to study completion, an average of 1 year.
Overall survival (OS) | From screening period up to study completion, an average of 1 year.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Sichuan Cancer Hospital, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: Undecided